CLINICAL TRIAL: NCT06064292
Title: Inspiratory Muscle Training in Adults With Cerebral Palsy: Long Term Effects. A Double-blind Randomised Controlled Trial
Brief Title: Long Term Effects of Inspiratory Muscle Training in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, CARLOS MARTIN SANCHEZ, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21032023
Record Dates: First submitted 2023-09-21; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Aging; Cerebral Palsy; Muscle Weakness; Older People--Abuse of; Physical Inactivity; Respiratory Tract Problem
MeSH Terms: conditions — Cerebral Palsy; Muscle Weakness; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: . The professional that collected the data and the participants were unaware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The High Intensity Training Group (HIT) (Experimental): The High Intensity Training Group (HIT) received IMT at 40% of Maximum Inspiratory Pressure (MIP), the training load was set each 2 weeks to keep 40% of MIP.
  Interventions: Device: INSPIRATORY MUSCLE TRAINING
- The Low Intensity Training Group (LIT) (Experimental): The Low Intensity Training Group (LIT) received IMT at 20% of MIP, following the same rules as HIT.
  Interventions: Device: INSPIRATORY MUSCLE TRAINING

INTERVENTIONS:
Device: INSPIRATORY MUSCLE TRAINING — After finishing the 8-week intervention period with IMT, CP patients stopped training with IMT and continued with their daily normal activities. During the following 24 weeks (without IMT), three evaluations of the respiratory parameters analyzed in the trial were made (MIP, MEP, FEV1, PEF). The first evaluation was made 4 weeks after the intervention was completed, the second 12 weeks and the third 24 weeks after finishing IMT.

SUMMARY:
Background: Respiratory disease is one of the main causes of morbidity and mortality in adults with cerebral palsy (CP). Adequate pulmonary function is essential to prevent these health problems, however respiratory muscle training has not yet been studied in CP patients. The main objective of the study was to investigate the maintenance over time of improvements in respiratory parameters achieved with inspiratory muscle training (IMT).

Methods: This was a controlled, randomised, double-blind trial and with allocation concealment performed on 27 institutionalized CP patients randomly distributed in 2 groups, "high intensity training group" (HIT) and "low intensity training group" (LIT). Participants followed a specific IMT program for 8 weeks, HIT workload was 40% of maximum inspiratory pressure (MIP) and LIT workload was 20% MIP. Once finished 8-week training period, CP patients continued their daily activities. Respiratory muscle strength and pulmonary function were measured pre-IMT, post-IMT, 4, 12 and 24 weeks after finishing IMT.

DETAILED DESCRIPTION:
Study design The study was a controlled, randomised, double-blind trial and with allocation concealment. The Bioethics Committee of the University of Salamanca affirms that the study meets ethical requirements for its execution (registry number 678)

Participants Institutionalized adults with CP aged between 35 and 64 years were included in the study, they were all members of ASPACE Salamanca. 38 patients with CP were selected to participate in the study. 27 participants were voluntarily recruited to participate in respiratory training and randomly distributed in the High Intensity Training Group (HIT) or Low Intensity Training Group (LIT).

Exclusion criteria: the presence of a respiratory disease in the previous month, inability to understand assessment tests or intervention or hemodynamic alterations (heart rate > 150 beats per minute (bpm), systolic blood pressure > 140 millimeters mercury (mmHg) or diastolic blood pressure > 90 mmHg).

The sample size was established by sampling calculation done from collected during a pilot study with 10 volunteers, which determined a minimum of 10 patients for each group to perceive differences of 12 cmH2O for MIP, power of 80%, security of 95%.

Procedures and Measures of Outcomes Elderly people with cerebral palsy were randomly allocated, via computerized random assignment, to either a high intensity intervention group or a low intensity intervention group. The professional that collected the data and the participants were unaware of group assignment. Before (pre-intervention) and after (post-intervention) inspiratory muscle training, respiratory muscle strength and pulmonary function were evaluated. Once the intervention period phase ended, 3 more evaluations of the same parameters were mare, the first at 4 weeks, the second at 12 weeks and the third at 24 weeks after finishing IMT.

Primary outcome The primary outcome was respiratory muscle strength, measured pre-IMT, post-IMT and 4, 12 and 24 weeks after finishing IMT intervention. It was evaluated through maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) using a pressure measurer (Elka PM-15, Laboliser, S.A., Barcelona, Spain), from residual volume and total lung capacity, severally. Each measure was expressed in millibars and turned into centimeter of water, reference unit, (cm H2O) (1 mbar = 1.01973 cm H2O), according to recommendations of the American Thoracic Society/European Respiratory Society (ATS / ERS) [24]. Each test was repeated 3 times or until 2 valid results were obtained (difference less than 5%). A rest time of 1 minute was respected between efforts to prevent short-term respiratory muscle fatigue. The highest value was selected. MIP was evaluated every 2 weeks to graduate the load of the device training.

Secondary outcome The secondary outcome was pulmonary function, measured pre-IMT, post-IMT and 4, 12 and 24 weeks after finishing IMT intervention. The data collected were forced expiratory volume in 1 second (FEV1) and peak expiratory flow (PEF). It was measured using the peak flow device (Asma-1, Vitalograph Ltd, Buckingham, England) that expresses the results of FEV1 in liters (L) and PEF in liters per minute (L/min), according to the guidelines of the ATS/ERS.

Experimental Protocol Inspiratory muscle training was carried out with a pressure threshold device (Treshold IMT, Philips-Respironics, Pittsburg, PA, USA). Threshold IMT provides consistent and specific pressure for inspiratory muscle strength and endurance training, regardless of how quickly or slowly patients breathe. This device incorporates a flow-independent one-way valve to ensure consistent resistance and features an adjustable specific pressure setting (in cm H2O) to be set by a healthcare professional. When patients inhale through Threshold IMT, a spring-loaded valve provides resistance. Before training began, the participants and primary caregivers completed one-session familiarization with a specialist to learn how to operate the device.

Adult people with cerebral palsy carried out the training program for 8 weeks, 1 session every day, 5 days a week. The participants performed 10 series of 1 minute with 1-minute rest between them.

The High Intensity Training Group (HIT) received IMT at 40% of MIP, the training load was set each 2 weeks to keep 40% of MIP. The Low Intensity Training Group (LIT) received IMT at 20% of MIP, following the same rules as HIT.

The training protocols of the two groups were developed by a specialist in respiratory therapy and all sessions with IMT were supervised by their main caregiver, therefore adherence to the program was controlled, as well as possible unwanted effects (increased fatigue, breathing problems, dizziness or sickness).

During the intervention period, both groups continued with their usual activity, receiving physiotherapy treatment for 45 minutes per day, 2 days per week. No participants received any other treatments.

After finishing the 8-week intervention period with IMT, CP patients stopped training with IMT and continued with their daily normal activities. During the following 24 weeks (without IMT), three evaluations of the respiratory parameters analyzed in the trial were made (MIP, MEP, FEV1, PEF). The first evaluation was made 4 weeks after the intervention was completed, the second 12 weeks and the third 24 weeks after finishing IMT.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized adults with cerebral palsy

Exclusion Criteria:

* The presence of a respiratory disease in the previous month
* Inability to understand assessment tests or intervention
* Hemodynamic alterations (heart rate > 150 beats per minute (bpm), systolic blood pressure > 140 millimeters mercury (mmHg) or diastolic blood pressure > 90 mmHg).

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle strength | 8 weeks.
  Maximum inspiratory pressure (MIP), unit of measure, Centimeters of water (cmH2O).

SECONDARY OUTCOMES:
Expiratory muscle strength | 8 WEEKS
  Maximum expiratory pressure (MEP), unit of measure, Centimeters of water (cmH2O).
Respiratory volume | 8 Weeks
  Forced expiratory volume in the first second (FEV1), unit of measure, liters (L).
Respiratory flow | 8 weeks.
  Peak expiratory flow (PEF), unit of measure, liters per minute (L/MIN).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Martin Sanchez, PhD, Principal Investigator — University of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No